CLINICAL TRIAL: NCT05636241
Title: The Effect of Whole Body Vibration on Walking Parameters in Children With Cerebral Palsy
Brief Title: Whole Body Vibration in Children With Cerebral Palsy
Acronym: CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Eda Ozge OKUR, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WBWinCP
Record Dates: First submitted 2022-10-28; First posted 2022-12-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Palsy; Spastic
Keywords: cerebral palsy; whole body vibration; gait; balance
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The participants in the control group will be attended to conventional physiotherapy program.
  Interventions: Other: conventional physiotherapy program
- study group (Experimental): The participants in the study group will be attended to whole body vibration training program.
  Interventions: Other: whole body vibration training program

INTERVENTIONS:
Other: conventional physiotherapy program — The conventional physiotherapy program consists of stretching exercises for lower extremities, strength exercises for core, upper, and lower extremity muscles, sit to stand exercises, and balance exercises.
  Arms: control group
Other: whole body vibration training program — The whole body vibration training program sessions consisted of three 3-min bouts of vibration of 20 Hz and a peak-to-peak amplitude of 2mm with a 3-min rest in between, in addition to conventional physiotherapy exercises for children with cerebral palsy.
  Arms: study group

SUMMARY:
Some positive effects of whole body vibration applications in reducing spasticity, improving walking ability, and increasing walking speed have been reported in children with CP, but the evidence is not strong enough. Therefore, this study was planned to evaluate the effect of whole body vibration treatment on spasticity, gait, balance, and motor performance in children with spastic CP. This study hypothesis that whole body vibration provides an additive improvement on spasticity, balance, gait and motor performance.

DETAILED DESCRIPTION:
Participants will be evaluate at baseline, after the conventional physiotherapy program, and after whole body vibration training program. During this period, the participants who were recruited whole body vibration training program, whole body vibration will be applied in addition to conventional physiotherapy sessions comprised 45 min, 2 days a week, during 8 week.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with spastic diplegic CP in GMFCS levels I and II, CFCS level I and MACS levels I and II
* Aged 6-17 years
* Ability to cooperate with the evaluations
* Walking independently with or without an orthosis (without any support)

Exclusion Criteria:

* Having a recent injury affecting the lower extremities
* Having undergone any surgery or Botulinuim Toxin application within the last six months
* Having severe cardiopulmonary or systemic problems
* Having uncontrolled seizures, visual or hearing problems preventing the evaluations

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Spatiotemporal parameters of gait will be evaluated with the Zebris™ FDM-2 gait analysis platform. | Change from baseline step length at 2 months.
  Gait analysis will be performed without any shoes and assistive devices. Walking evaluation on the gait platform will be limited to 1 minute. Obtained data about step length will be collected as centimeters from the entire 1-minute walk will use for analysis.
Spatiotemporal parameters of gait will be evaluated with the Zebris™ FDM-2 gait analysis platform. | Change from baseline stride length at 2 months.
  Gait analysis will be performed without any shoes and assistive devices. Walking evaluation on the gait platform will be limited to 1 minute. Obtained data about stride length will be collected as centimeters from the entire 1-minute walk will use for analysis.
Spatiotemporal parameters of gait will be evaluated with the Zebris™ FDM-2 gait analysis platform. | Change from baseline step width at 2 months.
  Gait analysis will be performed without any shoes and assistive devices. Walking evaluation on the gait platform will be limited to 1 minute. Obtained data about step width will be collected as centimeters from the entire 1-minute walk will use for analysis.
Spatiotemporal parameters of gait will be evaluated with the Zebris™ FDM-2 gait analysis platform. | Change from baseline step time at 2 months.
  Gait analysis will be performed without any shoes and assistive devices. Walking evaluation on the gait platform will be limited to 1 minute. Obtained dataabout step time will be collected as seconds from the entire 1-minute walk will use for analysis.
Spatiotemporal parameters of gait will be evaluated with the Zebris™ FDM-2 gait analysis platform. | Change from baseline cadance at 2 months.
  Gait analysis will be performed without any shoes and assistive devices. Walking evaluation on the gait platform will be limited to 1 minute. Obtained data about cadence will be collected as counts of steps from the entire 1-minute walk will use for analysis.
Spatiotemporal parameters of gait will be evaluated with the Zebris™ FDM-2 gait analysis platform. | Change from baseline velocity at 2 months.
  Gait analysis will be performed without any shoes and assistive devices. Walking evaluation on the gait platform will be limited to 1 minute. Obtained data about velocity will be collected as meters/seconds from the entire 1-minute walk will use for analysis.

SECONDARY OUTCOMES:
The Pediatric Balance Scale will be used to measure functional balance of the participants. | Change from baseline score at 2 months.
  Scale consist of 14-item. The highest score that can be obtained from the scale is 56. Highest scores shows better balance skills.

OTHER OUTCOMES:
Spasticity level of the participants will be measure with Modified Ashworth Scale. | Change from baseline score at 2 months.
  Muscle tone will be evaluated using the Modified Ashworth Scale from the right and left elbow flexors, forearm pronators, knee flexors, ankle plantar flexors, and hip adductors. The possible scores ranged from 0-4 for each movement, and lower scores indicate better outcome and higher scores indicate worse outcome.
Functional mobility of the participants will be measure with 1-min walk test. | Change from baseline distance at 2 months.
  Participants will be tested with their usual walking aids, orthoses and shoes. Before the test, a trial test will be performed. After 5 minutes resting period, the participant will be asked to walk as fast as possible without running on the 20 meter oval track during 1 minute. When the time is over, the distance the participant has walked will be measured in meters and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Ozge Okur, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- KMSU, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han YG, Lee SW, Yun CK. The immediate influence of various whole-body vibration frequency on balance and walking ability in children with cerebral palsy: a pilot study. J Exerc Rehabil. 2019 Aug 28;15(4):597-602. doi: 10.12965/jer.1938318.159. eCollection 2019 Aug. PMID 31523683